CLINICAL TRIAL: NCT04589039
Title: Post-Marketing Surveillance (Usage Results Study) of Niraparib in the Treatment of Adult Patients for Approved Indications in South Korea
Brief Title: A Study for Post-Marketing Surveillance of Niraparib in the Treatment of Adult Participants for Approved Indications in South Korea
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: Niraparib-5001; U1111-1257-0180 (Registry Identifier: WHO)
Record Dates: First submitted 2020-10-13; First posted 2020-10-19 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Ovarian Neoplasms
Keywords: Drug Therapy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants with Ovarian Cancer: Participants diagnosed with ovarian cancer (including fallopian tube or primary peritoneal cancer) who have been prescribed with niraparib for the first time in a real-world setting, and who are in a complete or partial response to first-line platinum-based chemotherapy or who had complete or partial response to 2 or more line of platinum-based chemotherapy or who have been treated with 3 or more prior chemotherapy regimens with either breast cancer susceptibility gene (BRCA) mutation (irrespective of platinum sensitivity) or platinum-sensitive homologous recombination deficiency (HRD) positive will be observed prospectively over 24-month period, or until treatment discontinuation, or until end of study, which occurs first.

SUMMARY:
The purpose of this study is to estimate the cumulative incidence of all adverse events (AEs), including serious adverse events (SAEs), adverse event of special interest (AESI), among participants who have been administered niraparib as per the approved indications.

DETAILED DESCRIPTION:
This is a long-term prospective, observational post-marketing surveillance study of niraparib in participants with ovarian cancer (including fallopian tube, or primary peritoneal cancer) who are in complete or partial response to first-line platinum-based chemotherapy or who had complete or partial response to 2 or more lines of platinum-based chemotherapy or who have been treated with 3 or more prior chemotherapy regimens with either: BRCA mutation irrespective of platinum sensitivity; or platinum-sensitive HRD positive. The study will assess the safety and effectiveness of niraparib for its approved indication with real-world setting in South Korea.

The study will enroll approximately 600 participants. The data will be collected prospectively at the study sites will be recorded into electronic case report forms (e-CRFs). All the participants will be assigned to a single observational cohort:

• Participants With Ovarian Cancer

The multi-center study will be conducted in South Korea. Data collection will be based on routinely scheduled and emergency visits during a 24-month surveillance period or until end of the study whichever occurs first after drug administration. The overall duration of the study will be approximately 6 years.

ELIGIBILITY:
Inclusion Criteria:

1. Monotherapy for the maintenance treatment of adult participants with ovarian, fallopian tube, or primary peritoneal cancer who are in a complete or partial response to first-line platinum-based chemotherapy.
2. Monotherapy for the maintenance treatment of adult participants with recurrent high-grade serous ovarian cancer (including fallopian tube, or primary peritoneal cancer) who are in a complete or partial response to 2 or more lines of platinum-based chemotherapy.
3. Monotherapy treatment of adult participants with recurrent ovarian, fallopian tube or primary peritoneal cancer who have been treated with three or more prior chemotherapy regimens with either a) BRCA mutation (irrespective of platinum sensitivity) or b) platinum-sensitive HRD positive.

Exclusion Criteria:

1. Treated with niraparib outside of the locally approved label in Korea.
2. Niraparib is contraindicated as per product label.
3. Participating in other clinical trials of cancer treatment.

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who have been prescribed niraparib for the first time in a real-world setting as a monotherapy treatment for participants with recurrent ovarian, fallopian tube or primary peritoneal cancer.
Sampling Method: Non-Probability Sample
Enrollment: 662 (Actual)
Dates: Start 2020-03-16 (Actual); Primary Completion 2024-09-11 (Actual); Study Completion 2024-09-11 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with AEs, SAEs, and AESIs | Baseline up to 24 months

SECONDARY OUTCOMES:
Time-to-Treatment Discontinuation (TTD) | From the date of first dose administration until discontinuation or death due to any cause whichever occurs first (up to 24 months)
  TTD is defined as the time interval from the date of initiation of treatment until discontinuation of treatment, or death due to any cause, whichever occurs first. Participants who have not discontinued treatment, or died, will be censored at the last known time that the participant was on treatment.
Progression Free Survival (PFS) | From the date of first dose administration until disease progression or death due to any cause whichever occurs first (up to 24 months)
  PFS is defined as the time interval from the date of initiation of treatment until objectively documented disease progression, or death due to any cause, whichever occurs first. Participants who do not have disease progression, or have not died, will be censored at the last known time that the participant was progression-free. Progressive disease (PD) is defined as at least a 20 percent (%) increase in the sum of the longest diameter (LD) of lesions, taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. The determination of disease progression will be at the Investigators discretion per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Inje University Haeundae Paik Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/